CLINICAL TRIAL: NCT04125888
Title: Impact of AIT on Allergic Rhinitis and Asthma Using Real World Evidence
Brief Title: Impact of AIT on Allergic Rhinitis and Asthma
Status: Completed | Type: Observational
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NI-X-04
Record Dates: First submitted 2019-10-04; First posted 2019-10-14 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Allergy; Respiratory Disease
MeSH Terms: conditions — Hypersensitivity; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AIT Cohort: Allergic rhinitis patients with and without asthma treated with AIT
  Interventions: Drug: Allergy immunotherapy (AIT)
- Control Cohort: Allergic rhinitis patients with and without asthma not treated with AIT

INTERVENTIONS:
Drug: Allergy immunotherapy (AIT) — Immunotherapy for different types of allergies
  Groups: AIT Cohort

SUMMARY:
The study will assess the effectiveness of AIT treatment in real clinical practice in Germany.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) affects 23-30% of the European population and is associated with a major burden on public health. AR and asthma frequently coexist, and may both be caused by allergen exposure. While the efficacy of AIT, i.e. reduce symptoms and medication use in patients with AR and asthma, has been demonstrated in several randomized clinical trials, little is known about the use and effectiveness of AIT in real world clinical practice.

This study is a retrospective database study that uses real-world data from Germany. The study population consists of AR patients with and without asthma treated with AIT and matched controls not treated with AIT. Information about the patients and treatments will be obtained from the 'BKK German Sickness Fund Database' from 2007 until 2017.

ELIGIBILITY:
Inclusion Criteria for the AIT cohort:

* At least two index-AIT prescriptions during the first FU-year
* At least one confirmed AR diagnosis during the study period
* Continuous enrollment (no gaps in insurance time-defined by days) for 12 months before the index event (in the pre-index period)
* Continuous enrollment (no gaps in insurance time-defined by days) for at least 12 months after the index event (in the post-index period)

Inclusion Criteria for the Control Cohort:

- For the control groups, the same inclusion criteria will apply, with the exception of inclusion criterion 1, i.e. controls have not received AIT before baseline.

Exclusion Criteria:

- AIT prescription 12 months before the index event (in the pre-index period) for the AIT treatment group

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Allergic rhinitis patients with and without asthma
Sampling Method: Probability Sample
Enrollment: 92048 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Allergic rhinitis medication use | From pre-index year to follow-up year(s), assessed from 2007 and up to 2017
  Number of patients with an AR prescription and number of prescriptions by drug class

SECONDARY OUTCOMES:
Asthma medication use | From pre-index to follow-up year(s), assessed from 2007 and up to 2017
  Number of patients with an asthma prescription and number of prescriptions by drug class
Change in asthma disease severity | From pre-index to follow-up year(s), assessed from 2007 and up to 2017
  Change in asthma disease severity assessed by asthma diagnoses, asthma medication use and severe asthma exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Romano, PharmD, MBA, MSc, Study Director — ALK Abelló
Locations (1):
- ALK Abelló, Hørsholm, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fritzsching B, Contoli M, Porsbjerg C, Buchs S, Larsen JR, Elliott L, Rodriguez MR, Freemantle N. Long-term real-world effectiveness of allergy immunotherapy in patients with allergic rhinitis and asthma: Results from the REACT study, a retrospective cohort study. Lancet Reg Health Eur. 2021 Nov 30;13:100275. doi: 10.1016/j.lanepe.2021.100275. eCollection 2022 Feb. PMID 34901915